CLINICAL TRIAL: NCT05757193
Title: Ketone Pharmacokinetic Study in Heart Failure With Reduced Ejection Fraction
Brief Title: Ketone Pharmacokinetic Study in HFrEF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00111723; K23HL161348 (NIH)
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: DeltaG; ketone ester; metabolites; metabolomics; ketoacidosis
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: Participants stratified based on use of background use of SGLT2 inhibitors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 250 mg/kg ketone ester (Experimental): The first 5 patients within each SGLT2i stratum will receive ketone ester as (R)-3-hydroxybutyl (R)-3-hydroxybutyrate at 250 mg/kg.
  Interventions: Dietary Supplement: DeltaG (250 mg/kg)
- 500 mg/kg ketone ester (Experimental): The second 5 patients within each SGLT2i stratum will receive ketone ester as (R)-3-hydroxybutyl (R)-3-hydroxybutyrate at 500 mg/kg.
  Interventions: Dietary Supplement: DeltaG (500 mg/kg)

INTERVENTIONS:
Dietary Supplement: DeltaG (250 mg/kg) — 250 mg/kg of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate
  Arms: 250 mg/kg ketone ester
Dietary Supplement: DeltaG (500 mg/kg) — 500 mg/kg of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate
  Arms: 500 mg/kg ketone ester

SUMMARY:
The purpose of this study is to test whether an over-the-counter ketone ester drink is well tolerated in people with heart failure on, and not on, a heart failure medication class called SGLT2 inhibitors. The research team is trying to determine the safest dose of Delta G. The study has a single visit. Participants will be served a light breakfast with the study drink, a physical exam will be conducted, and the study team will obtain information about demographics and medical history. The study team will draw blood intravenously up to eight times over the course of the half-day visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HFrEF (ejection fraction<=45%)
* Systolic blood pressure greater >=90 mmHg

Exclusion Criteria:

* Intentional ketogenic (high fat, low carbohydrate) diet (must be off ketogenic diet for >7 days prior to visit)
* Significant liver disease (cirrhosis) or alcohol abuse disorder (>14 drinks/week).
* Unique cardiomyopathies: infiltrative/hypertrophic cardiomyopathy, pericardial disease, or other cardiomyopathies that in the investigator's opinion have unique treatment options that would be less likely to be affected by ketone therapy.
* Estimated glomerular filtration rate<25 mL/min/1.73 m2 as the most recent value in the last year.
* Type 1 diabetes mellitus
* Use of ventricular assist device, history of heart transplant, or use of continuous inotropes
* Pregnant women. Due to unknown affects of nutritional ketosis in pregnant women, pregnancy will be an exclusion. Accordingly, women of childbearing age with a menstrual cycle within the past year will be asked to submit a urine specimen for pregnancy testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senthil Selvaraj, MD, MSTR, MA, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selvaraj S, Kwee LC, Thompson EJ, He M, Hornik CP, Devore AD, Patel CB, Mentz RJ, Fudim M, Taylor L, Milosovic S, Hurdle M, Cade WT, Ilkayeva O, Muehlbauer MJ, Newgard CB, Kelly DP, Zamani P, Margulies KB, Shah SH. Metabolic and Pharmacokinetic Profiling of a Ketone Ester by Background SGLT2 Inhibitor Therapy in HFrEF. JACC Basic Transl Sci. 2025 Mar;10(3):290-303. doi: 10.1016/j.jacbts.2024.10.014. Epub 2024 Nov 15. PMID 40139871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited within the Duke University Health System.
Groups:
- 250 mg/kg Ketone Ester: Participants received ketone ester as (R)-3-hydroxybutyl (R)-3-hydroxybutyrate at 250 mg/kg.
  DeltaG (250 mg/kg): 250 mg/kg of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate
- 500 mg/kg Ketone Ester: Participants received ketone ester as (R)-3-hydroxybutyl (R)-3-hydroxybutyrate at 500 mg/kg.
  DeltaG (500 mg/kg): 500 mg/kg of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate
Period: Overall Study
Arm/Group | 250 mg/kg Ketone Ester | 500 mg/kg Ketone Ester
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 250 mg/kg Ketone Ester | 500 mg/kg Ketone Ester | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.1) | 65.0 (9.0) | 64.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Venous pH Measured Via Peripheral Blood
Description: The pH scale ranges from 0 to 14, with 7 being neutral. Each number on the pH scale represents a ten-fold change in the acidity or basicity of a solution.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | 250 mg/kg Ketone Ester | 500 mg/kg Ketone Ester
Number analyzed (Participants) | 10 | 10
unitless | 7.30 (0.04) | 7.28 (0.04)

2. Primary Outcome: Glucose Level Measured Via Peripheral Blood
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 250 mg/kg Ketone Ester | 500 mg/kg Ketone Ester
Number analyzed (Participants) | 10 | 10
mg/dL | 136 (70) | 101 (45)

3. Primary Outcome: Systolic Blood Pressure
Description: Taken by blood pressure cuff on the arm
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 250 mg/kg Ketone Ester | 500 mg/kg Ketone Ester
Number analyzed (Participants) | 10 | 10
mmHg | 108 (12) | 110 (15)

4. Primary Outcome: Beta-hydroxybutyrate (BHB) Level Measured Via Peripheral Blood
Description: BHB is a chemical that is made by the body. It provides energy when not enough carbohydrates or sugars have been eaten.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: millimolar
Arm/Group | 250 mg/kg Ketone Ester | 500 mg/kg Ketone Ester
Number analyzed (Participants) | 10 | 9
millimolar | 1.88 (0.30) | 2.78 (0.54)

ADVERSE EVENTS:
Time Frame: Reported prior to the end of the study visit, up to 4 hours after ketone ester ingestion.
Arm/Group | 250 mg/kg Ketone Ester | 500 mg/kg Ketone Ester
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg/kg Ketone Ester (N=10) | 500 mg/kg Ketone Ester (N=10)
Headache (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT05757193/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT05757193/ICF_000.pdf